CLINICAL TRIAL: NCT07154511
Title: Phase 2 Trial of Tributyrin in People With Parkinson's Disease and Cognitive Impairments
Acronym: BUTTER2
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prabesh Kanel (Other)
Collaborators: Farmer Family Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Prabesh Kanel, Research Assistant Professor of Radiology, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00270219
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease; Parkinson Disease Dementia
Keywords: short chain fatty acid; butyrate; tributyrin; functional neuroimaging
MeSH Terms: conditions — Parkinson Disease | interventions — tributyrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tributyrin Supplementation (Experimental): Participants will take 500mg TID tributyrin supplement for 90 days +/- 7 days.
  Interventions: Drug: Tributyrin
- Placebo (Placebo Comparator): Participants will take 500mg placebo for 90 days +/- 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tributyrin — Post-biotic short chain fatty acid dietary supplement. Participants will take 500mg TID tributyrin supplement for 90 days +/- 7 days.
  Arms: Tributyrin Supplementation
Drug: Placebo — Participants will take 500mg TID placebo for 90 days +/- 7 days.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if taking a tributyrin supplement works to improve memory and thinking and walking and balance in adults with Parkinson disease Parkinson disease dementia. It will also learn about the safety of tributyrin supplementation. The main questions it aims to answer are:

1. Does tributyrin improve memory/thinking test scores and walking/balance ability?
2. What medical problems do participants have when taking tributyrin?

Researchers will compare tributyrin to a placebo (a look-alike substance that contains no drug) to see if tributyrin works to treat Parkinson disease symptoms.

Participants will:

1. Take tributyrin 3 times a day for 80-100 days
2. Complete motor and cognitive testing at the clinic before and after the supplementation period
3. Complete brain imaging (MRI scans and PET scans) before and after the supplementation period.

DETAILED DESCRIPTION:
Changes in cognition, progressing usually to dementia, are common features of Parkinson disease (PD). These debilitating impairments respond poorly to current anti-dementia treatments and call for novel strategies. Short chain fatty acids (SFCA), in particular butyric acid (BA), are naturally present in the colon as a bacterial product of dietary fiber fermentation. There is renewed interest in SCFAs because of their potential as alternative substrates in brain metabolism, their role in the gut-brain axis, and emerging evidence that interventions promoting SCFA benefit patients with neurodegenerative disorders. Convergent evidence suggests that SFCAs may ameliorate metabolic defects secondary to mitochondrial abnormalities in PD. In addition, the gut-brain axis represents a bidirectional communication complex system involving the vagal and sympathetic nerves and humoral systems. Effects of SCFA on the brain may be indirect and/or direct. For example, fiber-induced SCFA production in the colon may result in vagal nerve-mediated changes affecting the brain. Blood and brain levels of fiber-induced SCFA are naturally very low. SCFAs can be directly administered orally, resulting in higher portal vein and systemic plasma levels that may more potently affect brain functions. Oral butyrate supplementation, however, suffers from several limitations as plasma levels are low because of rapid metabolism. In contrast, tributyrin (the triglyceride of BA) is rapidly absorbed and chemically stable in plasma, diffuses through biological membranes and is metabolized by intracellular lipases, releasing therapeutically effective BA over time directly within cells. We previously generated target engagement data showing that oral tributyrin, 500 mg three times per day (tid) po, is well tolerated and improves cognition. We also conducted the first [11C]butyrate positron emission tomography (PET) study, demonstrating that tributyrin has direct brain effects, particularly in regions relevant to cognitive functions. Significant systemic anti-inflammatory effects were also observed. A limitation of our preliminary phase 1I target engagement study is the short duration (30 days) and lack of inclusion of people with PD with more severe cognitive impairments, such as dementia. The overarching goal of this project is to perform a parallel group, double-blinded, randomized placebo-controlled phase 2 clinical trial of tributyrin, 500 mg tid po for 90 days, to validate and extend these preliminary observations in a longer duration clinical trial in people with PD with mild cognitive impairment (PD-MCI) or Parkinson disease dementia (PDD). There is critical unmet clinical need to treat people currently affected with PD who have significant cognitive impairments. Our main hypothesis is that oral tributyrin supplementation will improve cognition as well as motor functions, including cognition-dependent postural instability and gait difficulties. Successful completion of this trial would set the stage for a major, multi-center phase III clinical trial aimed at ameliorating this particularly morbid feature of PD.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, age 45 years and over.
* Diagnosis of PD based on the United Kingdom Parkinson's Disease Society Brain Bank Diagnostic Research Criteria (Hughes et al., 1992) AND evidence of mild cognitive impairment (Litvan et al., 2012) OR Diagnosis of PDD (Emre et al., 2007).
* If taking cholinesterase inhibitors, benzodiazepines, memantine, or anti-psychotic medications, on a stable regimen as defined by no medication changes for these drugs in prior 4 weeks.

Exclusion Criteria:

* Evidence of atypical parkinsonism.
* Contra-indications to MR imaging including but not limited to pacemakers, aneurysm clips, intraocular metal, cochlear implant, or severe claustrophobia.
* Evidence of large vessel stroke or mass lesion on MRI.
* Regular use of typical anti-cholinergic drugs.
* Recent history of significant, uncontrolled GI disease such as GERD, colorectal cancer.
* Significant metabolic or uncontrolled medical comorbidity.
* Pregnant or nursing.
* Suicidal ideation, as indicated by a response of 2 or 3 on question 9 of the Beck Depression Inventory.
* Any other condition or criterion that would preclude safe and meaningful participation in the study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Single composite global cognitive z-score | Baseline and post-intervention (83-97 days after starting supplement)
  A global cognitive z-score derived from a neuropsychological battery including the California Verbal Learning Test (short- and long-term memory), Delis-Kaplan Executive Function System (verbal fluency via letter fluency test, executive function via Stroop and Trail Making Test Part 4), and Benton Judgment of Line Orientation Test (visuospatial cognition). Individual test scores are normatively z-scored with age- and sex-adjustment using data from 55 cognitively normal controls (Montreal Cognitive Assessment score > 25). All z-scores are aligned so that higher scores indicate better performance. Scores are averaged within domains and then across domains to compute the global cognitive z-score.
Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III Score | Baseline and post-intervention (83-97 days after starting supplement)
  Movement Disorder Society Unified Parkinson's Disease Rating Scale Part 3 (MDS-UPDRS part III) is the motor examination portion of the UPDRS evaluation. Scores range from 0-132, with higher scores indicating greater severity of motor symptoms.
Safety and tolerability of tributyrin | During and after 83-97 day supplementation period
  Safety and tolerability are assessed by monitoring the incidence, severity, and relationship of adverse events (AEs), serious adverse events (SAEs), and discontinuations due to AEs. AE information via biweekly phone-call monitoring, and during the post-intervention study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Prabesh Kanel, PhD, Principal Investigator — University of Michigan
Locations (1):
- Domino's Farms, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No